CLINICAL TRIAL: NCT05589181
Title: Safety and Efficacy of High Dose Buprenorphine Induction in Fentanyl Positive Emergency Department Patients
Brief Title: High Dose Buprenorphine (BUP) Induction in the Emergency Department (ED)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ethan Cowan, MD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2024002574; UG3DA056891 (NIH)
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: The design of Trial 1 and Trial 2 will be described separately. Trial 1 is a prospective test of the safety and tolerability of 32 mg of BUP as an induction dose (split dosing over 30-60 minutes with 4 hours of post-induction monitoring) with the recommended BUP induction dose (12mg, also split over 60 minutes). Trial 2 is a four-site pilot RCT (n=20x4) conducted in the ED, that will test the efficacy, safety and tolerability of the high BUP dose (selected in Trial 1) as an induction dose (split dosing over 30-60 min) compared to standard BUP induction dose (up to 12mg) also split over 30-60 min.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In trial 1 neither the investigator nor the participant will be blinded to group assignment. In Trial 2, participants, Investigators and site personnel with the exception of the investigational drug pharmacist will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buprenorphine Standard Dose (Active Comparator): The standard arm will receive an induction dose of 12mg of buprenorphine (BUP) split as 8mg at time=0 and 4mg at time=30-60 min.
  Interventions: Drug: Standard Buprenorphine Dose
- Buprenorphine High Dose (Experimental): The experimental arm tests the safety and tolerability of 32mg of BUP split as 16mg at time=0 and 16mg at time=30-60 min as an induction dose.
  Interventions: Drug: High Dose Buprenorphine

INTERVENTIONS:
Drug: High Dose Buprenorphine — 32mg of BUP split as 16mg at 0 minutes and 16mg at 30-60 min as an induction dose
  Arms: Buprenorphine High Dose
Drug: Standard Buprenorphine Dose — 12mg of buprenorphine (BUP) split as 8mg at 0 minutes and 4mg at time 30-60 min as an induction dose
  Arms: Buprenorphine Standard Dose

SUMMARY:
This project, involving two distinct clinical trials, tests whether induction to a higher than currently recommended buprenorphine (BUP) induction dose is safe and can improve the proportion of patients who engage in comprehensive addiction services within 7-day of induction.

Trial 1 is a head-to-head comparison of the safety, tolerability and feasibility of high dose BUP induction (32 mg). The study involves two cohorts, (1) a 12mg cohort (standard) to determine baseline data and (2) a 32 mg (high dose) cohort. If the 32mg is intolerable, a 24 mg dose may be evaluated. Trial 2 is a small pilot multicenter randomized, double blinded, clinical trial in 80 participants (randomized 1:1) that will provide preliminary information on efficacy with the primary outcome being engagement in comprehensive addiction treatment 7-days post BUP induction. In collaboration with National Institute on Drug Abuse (NIDA), the research team have determined that there must be a minimum increase in engagement in comprehensive addiction treatment of 15% at 7-days in the high dose induction group to justify a larger future clinical trial.

DETAILED DESCRIPTION:
The design of Trial 1 and Trial 2 will be described separately. Trial 1 is a prospective test of the safety and tolerability of 32 mg of BUP as an induction dose (split dosing over 30-60 minutes with 4 hours of post-induction monitoring) with the recommended BUP induction dose (12mg, also split over 60 minutes). Dosing for the 12 mg cohort is planned to be 8 mg at t=0 and 4 mg at 30-60 min. The dosing for the 32 mg cohort is planned to be 16 mg at t=0 and 16 mg at 30-60 min.

The frequency of unacceptable dose limiting toxicities is set at >10%. The study will therefore compare two cohorts of 10 participants, with the potential for 5 extra participants per cohort if 1 dose limiting toxicity is observed in the first 10 subjects in a cohort.

If there are two dose limiting toxicities (DLTs) in the 32mg cohort, that cohort will no longer recruit. A new, 24 mg high dose cohort will be formed. If the 24 mg cohort has 2 DLTs in either 1st 10 patients or when expanded to n=15, it will be concluded that no safe/tolerable high induction dose has been identified and trial 2 will not occur.

If the 12 mg (control) cohort has 2 DLTs, at n=15 the Data and Safety Monitoring Board (DSMB) will be consulted about enlarging the cohort size or other modifications.

Any participants in the 12 mg cohort who choose not to take their full assigned dose will be replaced to ensure the full cohort size. No more than 20% of participants in either 24 mg or 32 mg cohorts who choose not to take their full assigned dose can be replaced.

Trial 1 will only take place in the Emergency Department at Mount Sinai Beth Israel Study participants can only be enrolled if they are active ED patients and only on the day of their ED visits. Patients will be screened by trained research associates (RAs) with a screener that includes questions about illicit opioid use in the past 30 days embedded in a general health and substance use screener that also includes questions about safety, tobacco and alcohol use. The screener will contain questions regarding opioid use and non-medical use of prescription opioids. Potential study patients who report any opioid use in the past month will complete a 7-day recall of such use. If opioid use is reported during the past 7 days a brief (10 minute) structured diagnostic interview with questions on the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) criteria will be used to evaluate the presence of moderate/severe opioid use. Those who meet study criteria will be informed that they may qualify for the study and will be then asked to provide a urine sample. If the urine tests are positive for fentanyl, the patient indicates ability to provide contract information for 1 separate reliable contacts (in addition to their own) and the patient meets all eligibility criteria on the Patient Eligibility Summary form, informed consent will be obtained.

Patients who sign written informed consent will be enrolled in the study and assigned to a dose cohort (either 12 or 32mg). Assignment in Trial 1 is sequential, not randomized. Participants will receive their full dose over 30-60 minutes and be observed for a total of 4-hours in the ED from the time of their first BUP dose. At the time of discharge all participants will receive a prescription for BUP for 7-day (16mg per day), harm reduction counseling that includes the provision of a naloxone rescue kit and fentanyl test strips and a referral for out-patient addiction treatment within 7-days of the ED visit. After discharge, study participants will be followed-up daily for 7 days to assess daily drug use and opioid craving. At 7-days all participants will be asked to return to provide a urine drug screen and be assessed for engagement in comprehensive addiction treatment and healthcare utilization.

Trial 2 is a four-site pilot randomized controlled trial (RCT) (n=20x4) conducted in the ED, that will test the efficacy, safety and tolerability of the high BUP dose (selected in Trial 1) as an induction dose (split dosing over 30-60 min) compared standard BUP induction dose (up to 12mg) also split over 30-60 min. The four sites participating in the Trial 2 RCT are, (1) Mount Sinai Hospital Emergency Department, (2) Mount Sinai Beth Israel Emergency Department, (3) Barnes Jewish Hospital Emergency Department and (4) Rhode Island Hospital Emergency Department.

Eligibility, screening and enrollment procedures are identical to Trial 1. Eligible participants will be randomized 1:1 with stratification by site to receive either standard (12mg) or high dose BUP induction (determined from trial 1 but no more than 32mg). Participants and study personnel will be blinded to group assignment. All participants will be observed in the ED for a total of 4-hours from the time of their first BUP dose. At discharge. all participants will receive a prescription for BUP for 7-day (16mg per day), harm reduction counseling that includes the provision of a naloxone rescue kit and fentanyl test strips and a referral for out-patient addiction treatment within 7-days of the ED visit. Participants will be followed-up at 7 and 14-day to assess the primary outcome (engagement in comprehensive addiction treatment) and multiple secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study
* Treated in the ED during screening hours
* Meet DSM-5 diagnostic criteria for moderate to severe OUD
* Clinical Opioid Withdrawal Score (COWS) score ≥ 8
* Urine toxicology positive for fentanyl
* Able to speak English or Spanish sufficiently to understand study procedures

Exclusion Criteria:

* UDS positive for methadone.
* Be pregnant determined by urine human chorionic gonadotropin (uHCG) testing
* Have an unstable medical or psychiatric condition including suicidality requiring hospitalization
* Require ongoing opioids for pain management
* Be enrolled in formal addition treatment including by court order anytime within the last 30 days. Patients enrolled in formal addiction treatment not receiving Medications for Opioid Use Disorder (MOUD) are eligible
* Be a prisoner or in custody at the time of the index visit
* Have any pending legal status or pending legal action that could prohibit full participation in or compliance with study procedures.
* Unable to provide one additional point of contact other than themselves
* Unwilling to follow study procedures
* Have prior enrollment in the current study
* Have a known allergy or hypersensitivity to BUP
* Have been engaged in formal addiction treatment in the 30-days prior to the ED visit (this does not include addiction treatment or residential programs where MOUD is not given (e.g. behavioral counseling, abstinence programs, NA)
* Have received naloxone in the 60-minutes prior to the anticipated first transmucosal (TM) BUP administration
* Is undergoing concurrent treatment with another investigational agent or enrolment in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants engaged in comprehensive addiction treatment at 7-days post-ED induction | 7 days post-ED visit
  The proportion of participants engaged in comprehensive addiction treatment at 7 days post-ED induction as verified by participant and the addiction treatment program.

SECONDARY OUTCOMES:
Percentage of days with opioid abstinence (Trial 1) | at day 7
  Participants' percentage of days with opioid abstinence (defined as negative urine drug screen (UDS)) at day 7 (Trial 1)
Percentage of days with opioid use (Trial 1) | 7 days post-ED
  Participants' percentage of days with opioid use at Time-Line Follow Back (TLFB) over 7 days post induction (inclusive) (Trial 1)
Percentage of days with opioid use (Trial 2) | 30 days post-ED
  Participants' percentage of days with opioid use at Time-Line Follow Back (TLFB) over 30 days post induction (inclusive) (Trial 2)
Daily assessment of opioid use (Trial 1) | Days 1-7 after enrollment
  Participants' daily assessment of opioid use out of days over a 7-day period (Trial 1)
Change in number of times opioids used (Trial 1) | induction through 7 days
  Change in participants' number of times opioids were per day used from induction through 7 days follow-up assessment (Trial 1)
Change in number of times opioids used (Trial 2) | Baseline and follow-up assessment day 7
  Change in participants' number of times opioids were used from baseline to follow-up assessment day 7 (Trial 2)
Change in number of times opioids used (Trial 2) | Baseline and follow-up assessment day 30
  Change in participants' number of times opioids were used from baseline to follow-up assessment day 30 (Trial 2)
Proportion of participants with persistent nausea/vomiting during induction | at 240 minutes
  Proportion of participants with persistent nausea/vomiting during the induction visit requiring treatment.
Proportion of participants with a Pasero Opioid-induced Sedation Scale (POSS) score of 3 or higher | at 240 minutes
  Proportion of participants with a POSS score of 3 or higher at the conclusion of the induction visit 4-hour observation period. Higher score indicates more severe sedation.
  S=sleep, easy to arouse
  1. awake/alert
  2. slight drowsy/easy aroused
  3. Frequently drowsy, arousable, drifts off to sleep during conversation
  4. Somnolent, minimal or no response to verbal and physical stimulation
Proportion of participants with a Mini Mental Status Exam (MMSE) score indicating severe cognitive impairment | at 240 minutes
  Proportion of participants with a Mini Mental Status Exam (MMSE) indicating severe cognitive impairment at the conclusion of the induction visit 4-hour observation period. The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language). Full scale ranges from 0-30, with higher scores indicating better function.
Proportion of participants with precipitated or worsening withdrawal | up to 240 minutes
  Proportion of participants with precipitated or worsening withdrawal requiring continued treatment with ancillary medications during the induction visit.
Patient Satisfaction Survey | ED enrollment visit at 240 minutes
  Patient Satisfaction Survey is a 4-item questionnaire, each item scores 1-5, with total score range of 4-20. Higher scores would indicate a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Cowan, MD, MS, Principal Investigator — The Rutgers Addiction Research Center
Locations (1):
- Rutgers University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
  This study will share deidentified individual participant data that underlie the results that are reported. The data intended for broader use will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning upon acceptance for publication and ending 5 years following article publication.
Access Criteria: deidentified individual patient data (IPD) will be shared with researchers who provide a methodologically sound proposal for the purpose of achieving aims in the approved proposal. Proposals should be directed to ethan.cowan@mountsinai.org.